CLINICAL TRIAL: NCT07235488
Title: Effectiveness of Integrative Medical Treatment in Sudden Hearing Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH113-REC2-096
Record Dates: First submitted 2025-09-23; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Sudden Hearing Loss
Keywords: sudden hearing loss; acupuncture
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steroid therapy combined with acupuncture (Experimental): Western Medicine Treatment: During hospitalization, intravenous steroids were administered. After discharge, oral steroids were administered. For patients who did not respond well to treatment, intratympanic steroid injections were performed.
  Traditional Chinese Medicine Treatment: Acupuncture was performed once daily for 30 minutes at acupoints around the ear and upper limb on the same side as the affected ear. Six treatment sessions were performed in the first and second weeks, and two sessions were performed in the third and fourth weeks.
  Interventions: Device: Acupuncture
- Steroid therapy (Active Comparator): Western Medicine Treatment: During hospitalization, intravenous steroids were administered. After discharge, oral steroids were administered. For patients who did not respond well to treatment, intratympanic steroid injections were performed.
  Interventions: Drug: steroid therapy

INTERVENTIONS:
Device: Acupuncture — Treatment lasted four weeks, starting from the date of admission, and included both inpatient and outpatient care.
  Western Medicine Treatment : During hospitalization, intravenous steroids were administered. After discharge, oral steroids were administered. For patients who did not respond well to treatment, intratympanic steroid injections were performed.
  Traditional Chinese Medicine Treatment : Acupuncture was performed on peri-auricular and ipsilateral upper limb points, including Ermen (TE21), Tinggong (SI19), Tinghui (GB2), Shuaigu (GB8), Yifeng (TE17), Waiguan (TE5), and Zhongzhu (TE3). The treatment was administered once daily for 30 minutes. During the first and second weeks, a total of six sessions were carried out, followed by two sessions per week in the third and fourth weeks.
  Arms: Steroid therapy combined with acupuncture
Drug: steroid therapy — Treatment lasted four weeks, starting from the date of admission, and included both inpatient and outpatient care.
  Western Medicine Treatment : During hospitalization, intravenous steroids were administered. After discharge, oral steroids were administered. For patients who did not respond well to treatment, intratympanic steroid injections were performed.
  Arms: Steroid therapy

SUMMARY:
Sudden hearing loss is an emergency in otolaryngology that requires diagnosis and treatment as soon as possible. The golden treatment period is two weeks since the onset of the disease. However, modern medicine is still unable to fully understand the causes of the disease and in lack of corresponding effective treatments. Current therapies also have their own limitations and side effects. To find an effective and safe treatment, integrating with modern medicine and providing inpatient and outpatient medical care, is an important issue in clinical care. Traditional Chinese medicine has been clinically utilized for a long time with accumulated empirical experience and evidence for its efficacy. It can be used as an alternative therapeutic option for sudden hearing loss.

Being with a long period of clinical experience and evidence-based curative effect, acupuncture could be applied as an adjunctive treatment for the sudden hearing loss. Currently, this patient-centered, pragmatic clinical trial compares the effectiveness of using west medicine、combination of west medicine and traditional Chinese medicine. The aim of this study is to explore acceptable and beneficial strategy to reduce the clinical symptoms, to improve quality of life, and decrease medical expenses.

DETAILED DESCRIPTION:
Patients newly diagnosed with sudden deafness were randomly assigned in a 1:1 ratio to two groups: a Western medicine group and an integrated Chinese and Western medicine treatment group. Each group included 32 patients, for a total of 64 patients. Treatment lasted four weeks, starting from the date of admission, and included both inpatient and outpatient care.

Western Medicine Treatment: During hospitalization, intravenous steroids were administered. After discharge, oral steroids were administered. For patients who did not respond well to treatment, intratympanic steroid injections were performed.

Traditional Chinese Medicine Treatment: Acupuncture was performed once daily for 30 minutes at acupoints around the ear and upper limb on the same side as the affected ear. Six treatment sessions were performed in the first and second weeks, and two sessions were performed in the third and fourth weeks.

Primary Outcome: Pure-tone audiograms were performed at baseline, week 1, week 2, and week 4.

Secondary Outcome: Tinnitus Handicap Inventory and Dizziness Handicap Inventory were performed at baseline, week 1, week 2, and week 4. Blood biochemistry tests were performed at baseline. Adverse events were recorded throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, both male and female.
* Meeting the diagnostic criteria for sudden sensorineural hearing loss (SSNHL), defined as hearing loss of >30 dB affecting at least three consecutive frequencies within 3 days.
* Newly onset of hearing loss within 2 week.
* Fully understanding the purpose and procedures of the study and providing signed informed consent.

Exclusion Criteria:

* Central nervous system lesions such as vestibular schwannoma or traumatic brain injury.
* Middle ear or retrocochlear pathology.
* History of otologic surgery.
* Hemorrhagic disorders or coagulation abnormalities.
* Inability to cooperate with examinations due to dementia or psychiatric illness.
* Previous treatment for SSNHL on the same affected side within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Pure-tone audiograms | baseline, week 1, week 2, and week 4
  Changes from baseline to week 1, week 2, and week 4 of the intervention

SECONDARY OUTCOMES:
Tinnitus Handicap Inventory | baseline, week 1, week 2, and week 4
  Changes from baseline to week 1, week 2, and week 4 of intervention
Dizziness Handicap Inventory | baseline, week 1, week 2, and week 4
  Changes from baseline to week 1, week 2, and week 4 of intervention
Blood examination | baseline
  neutrophil-to-lymphocyte ratio (NLR)
Laboratory examination | baseline
  inflammatory cytokine test (IL-1β, IL-6, TNF-α)
Adverse events | baseline, week 1, week 2, and week 4
  Adverse events related to steroid or acupuncture therapy were recorded throughout the trial.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No